CLINICAL TRIAL: NCT04404062
Title: Serological and PCR Testing for SARS-CoV-2. A Prospective Study Assessing Infection, Immunity, and Asymptomatic Carriage of COVID-19
Brief Title: Serological and PCR Testing for COVID-19
Status: Recruiting | Type: Observational
Sponsor: Richmond Research Institute (Industry)
Collaborators: Richmond Pharmacology Limited (Industry)
Responsible Party: Sponsor
Organization: Richmond Pharmacology Limited (Industry)
Other Study IDs: C20010
Record Dates: First submitted 2020-05-22; First posted 2020-05-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Trial Participants: Male and female participants aged 5-70 years
  Interventions: Diagnostic Test: Membrane-based immunoassay kit; Diagnostic Test: Quantitative antibody Tests; Diagnostic Test: PCR Test

INTERVENTIONS:
Diagnostic Test: Membrane-based immunoassay kit — The kit is a qualitative membrane-based immunoassay to detect IgG and IgM antibodies to SARS-CoV-2 in whole blood, serum or plasma specimens. IgG and IgM detection components are separate allowing for differential detection of each antibody.
  Other Names: Covid-19 Rapid Test Kit
Diagnostic Test: Quantitative antibody Tests — Antibody titres will be measured from whole blood samples taken from volunteers.
  Other Names: Antibody titre
Diagnostic Test: PCR Test — PCR tests will be conducted on throat swabs taken from volunteers.

SUMMARY:
Richmond Research Institute (RRI) is applying existing and new COVID-19 PCR and antibody tests to help develop methodologies which provide fast and accurate results. Infection with coronavirus (SARS-CoV-2) is currently a worldwide pandemic and reliable testing for COVID-19 is crucial to understand who is infected and therefore a risk to others by spreading the infection. RRI are currently carrying out the following tests:

A. Using a membrane-based immunoassay to detect IgG and IgM antibodies to SARS-CoV-2 in whole blood, serum or plasma specimens helps to assess whether an individual has previously had the virus and is potentially immune

B. Polymerase Chain Reaction (PCR) testing using an established method to check for active SARS-CoV-2 infections.

C. Quantification of anti-SARS-CoV-2 IgG and IgM antibodies in whole blood samples.

The above tests are being used by RRI to follow infections (PCR) and immunity (IgG) in their workforce, as well as their families (including children) and visitors to their site.

Collecting this data allows the gathering of epidemiological data on SARS-CoV-2 including incidence, prevalence, information on asymptomatic carriers and efficacy of vaccination. Furthermore, identifying individuals that are infected with SARS-CoV-2 has great potential to improve health outcomes by allowing infected individuals to seek the correct medical treatment as well as self-isolate and reduce transmission.

DETAILED DESCRIPTION:
This is a screening study to measure symptomatic and asymptomatic carriage of SARS-CoV-2 in trial participants to help facilitate early detection of a second wave of SARS-CoV-2 infections. Specifically, this study aims to determine ; to assess the duration of immunity by assessing the number and speed at which trial participants were infected and cleared the virus with or without symptoms; and to determine the length of symptom onset in those with an active infection; levels of IgG antibodies by demographics (sex, age, ethnicity, and intensity of symptoms). Longitudinal assessment of antibody levels will additionally allow for assessment of the efficacy of any vaccines adminstered. This study also seeks to explore how many people are asymptomatic carriers. In addition, this study aims to help facilitate the development a quantitative laboratory reference test for antibodies (IgG).

By using multiple different tests, it can be determined if a person is currently infected with SARS-CoV-2 or whether they previously have been infected. This allows for the scanning of people with asymptomatic carriage of the virus, which is important to help reduce the spread of SARS-CoV-2 through contact with people unaware of infection.

Polymerase Chain Reaction (PCR) testing is routinely used to check for active SARS-CoV-2 infections. It measures whether viral RNA is present in an individual's system. All in-house PCR tests are verified by an independent laboratory to check for false positives.

Using a membrane-based immunoassay to detect IgG and IgM antibodies to SARS-CoV-2 in whole blood, serum or plasma specimens helps to assess whether an individual has previously had the virus and is potentially immune. IgG and IgM detection components are separate allowing for differential detection of each antibody.

To this date, 20904 PCR tests and 6848 antibody tests have been carried out in 2328 individuals, providing some interim data. Of the 20904 PCR tests, 17635 (84%) were negative and 132 (1%) were negative. Of the 6848 antibody tests, 706 (10%) were positive for IgG only, 64 (1%) were positive for IgM only, and 351 (5%) were positive for both IgG and IgM. 5710 (83%) tests were negative.

Of those individuals with a positive PCR test, 53% reported fever during the previous two months and 75% reported a loss of taste during the previous two months.

Interim results are shown in the medRxiv papers below:

https://www.medrxiv.org/content/10.1101/2020.12.08.20245894v2

https://www.medrxiv.org/content/10.1101/2021.04.09.21255200v1

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 5 to 70 years.
* An understanding, ability, and willingness to fully comply with the project procedures and restrictions.

Exclusion Criteria:

* Not applicable.

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants are individuals who are screened upon entry to the Richmond Pharmacology unit. These individuals may be employees of Richmond Pharmacology, volunteers for other concurrent studies, or members of the public.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2020-03-16 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Identification of carriers of SARS-CoV-2 | Through study completion, estimated 12 weeks
  To identify trial participants who are symptomatic or asymptomatic carriers of SARS-CoV-2 by comparing the results of a blood finger stick test and reference laboratory tests to PCR testing for acute infection

SECONDARY OUTCOMES:
Determination of the duration of immunity to SARS-CoV-2 | Through study completion, estimated 12 weeks
  To determine the duration of immunity of trial participants previously infected with SARS-CoV-2, measure differences in IgG antibodies by demographics including sex, ethnicity and age and investigate correlation between IgG antibody levels and intensity of symptoms
Development of a quantitative laboratory reference test for the measurement of SARS-CoV-2 | Through study completion, estimated 12 weeks
  Determination of the understanding of the quantity of IgG antibodies developed as a response to SARS-CoV-2 infection, and how these antibody levels decrease over time. Antibody titres will be measured in infected individuals, over multiple days and correlated with disease parameters. This will facilitate the development of a quantitative laboratory reference test for IgG antibodies
Exploration of SARS-CoV-2 epidemiology | Through study completion, estimated 12 weeks
  To help develop a quantitative laboratory reference test for antibodies (IgG) to gain an understanding of quantity of antibodies that people develop and how these decrease over time.

CONTACTS AND LOCATIONS:
Overall Officials: Jorg Taubel, MD, Principal Investigator — Richmond Pharmacology Limited
Locations (1):
- Richmond Pharmacology Ltd. 1a Newcomen St, London Bridge, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No